CLINICAL TRIAL: NCT03570008
Title: Preventing the Risk of Osteoporotic Fracture in Premenopausal Women by a Spa Residential Physical Activity Program
Acronym: ThermOs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Regional Council of Auvergne-Rhône-Alpes (Other); European Regional Development Fund (Other); Spa resort of Chaudes Aigues, 27 avenue Georges Pompidou, BP21, 15110 Chaudes Aigues, France (Unknown); Spa resort of Bourbon-Lancy, place d'Aligre 71140 Bourbon-Lancy, France (Unknown); Innovatherm (Industry); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHU-387; 2016-A02083-48 (Other: 2016-A02083-48)
Record Dates: First submitted 2018-03-26; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Osteoporotic Fracture
Keywords: prevention; bone; physical activity; spa bath; women
MeSH Terms: conditions — Osteoporotic Fractures; Motor Activity | interventions — Exercise

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sp-Ex (Experimental): a 9 days spa residential program including physical activity. 3 sessions of 10 minutes per day of physical exercise for bone health improvements supervised by a professional of adapted physical activity. Participants will benefit advices from national plan for physical activity and nutrition (NPPN)
  Interventions: Behavioral: 9 days spa residential program; Behavioral: 3 sessions of 10 minutes per day of physical exercise
- Sp-alone (Active Comparator): Participants will benefit a short term spa residential program of 9 days. In addition they will benefit advices from national plan for physical activity and nutrition (NPPN)
  Interventions: Behavioral: 9 days spa residential program
- Ex-alone (Active Comparator): Participants will benefit 3 sessions of 10 minutes per day of physical exercise for bone health improvements supervised by a professional of adapted physical activity. Participants will benefit advices from national plan for physical activity and nutrition (NPPN)
  Interventions: Behavioral: 3 sessions of 10 minutes per day of physical exercise

INTERVENTIONS:
Behavioral: 9 days spa residential program — After the inclusion visit, the participants will be involved in a short-term spa residential program of 9 days (Sp). The will be randomized into 3 groups of 30 participants:
  * Sp-Ex: spa residential program including physical activity
  * Sp-alone: spa residential program alone
  * Ex-alone: physical activity alone
  After the spa residential program, participants will undergo a one-year at-home follow-up. The participants will be required to complete the same program by themselves.
  A journal and an accelerometer-pedometer watch will record the weekly physical activity performed. Monitoring will be further monthly assessed by a health-care professional from the spa resorts.
  Arms: Sp-Ex; Sp-alone
Behavioral: 3 sessions of 10 minutes per day of physical exercise — After the inclusion visit, the participants will be involved in a short-term spa residential program of 9 days (Sp). The will be randomized into 3 groups of 30 participants:
  * Sp-Ex: spa residential program including physical activity
  * Sp-alone: spa residential program alone
  * Ex-alone: physical activity alone
  After the spa residential program, participants will undergo a one-year at-home follow-up. The participants will be required to complete the same program by themselves.
  A journal and an accelerometer-pedometer watch will record the weekly physical activity performed. Monitoring will be further monthly assessed by a health-care professional from the spa resorts.
  Arms: Ex-alone; Sp-Ex

SUMMARY:
Osteoporosis is an increasing public health problem. Involution of bone mass in women is due to a reduction in sensitivity of the bone to the mechanical stress due to the slow-down of the bone turnover after 35 years old. Osteoporosis is a silent disease combining a decrease in bone mass (quantity) and an impaired bone microarchitecture (quality) leading to an increased risk of fracture. Bone microarchitecture is an important element to be taken into account in assessing the bone properties, as demonstrated by numerous ex vivo studies.

Bone densitometry only identifies 50% of osteoporotic fractures. The other half of the fractures appears in osteopenic women. The measurement of bone mineral density is too limited to assess risk of fracture. Bone microarchitecture can be assessed through a peripheral quantitative computed tomography scan (computed tomography peripherical - pQCT). The microarchitecture data allow the calculation of bone strength index (BSI) and stress strength index (SSI) highly predictive of fracture risk. These qualitative determinants of bone fragility are the most relevant to evaluate effect of physical activity over a short period compared with bone mineral content and density, which requires several months of constraints. Biochemical markers of bone turnover, specifically those of bone resorption, are predictive of the risk of osteoporotic fracture.

Physical activity can reduce the risk of fracture up to 20-35% via direct effects on bone strength, at any age. However, response of bone varies with modalities of exercise. Repeated exercise produces greater bone adaptations than a single bout. Moreover, it has been well demonstrated since 1970 that bone responds to a dynamic stimulation, but not a static stimulation, with a dose response relationship. It has been confirmed in premenopausal women.

The effect of physical activity on microarchitectural bone parameters (porosity and density of cortical and trabecular) has not been investigated in primary prevention. This original study would highlight the effect of short-term specific physical activity on the prevention of bone fragility (qualitative) observed with age in premenopausal women.

The main hypothesis is that a spa residential program including physical activity will have greater benefits on bone cortical porosity than a spa residential program alone or physical activity alone, in premenopausal women.

DETAILED DESCRIPTION:
The ThermOs protocol was designed to provide a better understanding of the effect of physical activity on microarchitectural bone parameters (porosity and density of cortical and trabecular), in prevention of bone fragility among premenopausal women.

In the present protocol, parameters are measured on four occasions (baseline, 10 days, at 6 months and at 12 months).

Statistical analysis will be performed using Stata software (version 13; Stata-Corp, College Station, Tex., USA). All statistical tests will be two-sided and p<0.05 will be considered significant. After testing for normal distribution (Shapiro-Wilk test), data will be treated either by parametric or non-parametric analyses according to statistical assumptions.

Inter-groups comparisons will systematically be performed 1) without adjustment and 2) adjusting on factors liable to be biased between groups.

Analysis will be performed using anova or Kruskal-Wallis (KW) tests. When appropriate (p<0.05), a post-hoc test for multiple comparisons (Tukey-Kramer after anova and Dunn post KW) will be used. Linear regression (with logarithmic transformation if necessary) considering an adjustment on covariates fixed according to epidemiological relevance and observance to physical activity will complete the analysis. Relations between quantitative outcomes will be analyzed using correlation coefficients (Pearson or Spearman) and compared with Chi-squared or Fischer test. Longitudinal data will be treated using mixt-model analyses in order to treat fixed effects group, time and group x time interaction taking into account between and within participant variability.

ELIGIBILITY:
Inclusion Criteria:

* Women with regular cycles
* 40-50 years old
* Sedentary lifestyle
* stable body weight over the previous 6 months
* Normal weighted (BMI<30)
* written informed consent.
* Affiliated to French health care system (for France)

Exclusion Criteria:

* Menopausal women
* Regular physical activity > 4 hours / week of moderate or high intensities
* Participant refusal to participate
* Hepatic, renal, or psychiatric diseases, nor cardiovascular or endocrine diseases (thyroid diseases will be included)
* HIV infection
* Use of medications altering body weight, corticosteroids, Nonsteroidal anti-inflammatory drugs
* Use of medications influencing bone parameters such as bisphosphonate, other osteoporotic treatment therapy, or chemotherapy
* Regular alcohol consumption (>20g of alcohol per day)
* Restricted diet over the previous 6 months
* Deficit or supplementation in vitamin D
* Protected persons are not excluded

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Variation of bone cortical porosity in premenopausal women after the interventional phase. | at Baseline
  To evaluate the effectiveness of a spa residential program including physical activity (Sp-Ex) on bone cortical porosity compared with a spa residential program alone (Sp-alone) or physical activity alone (Ex-alone), in premenopausal women.
Variation of bone cortical porosity in premenopausal women | after 10 days
  To evaluate the effectiveness of a spa residential program including physical activity (Sp-Ex) on bone cortical porosity compared with a spa residential program alone (Sp-alone) or physical activity alone (Ex-alone), in premenopausal women.
Variation of bone cortical porosity in premenopausal women | after 6 months
  To evaluate the effectiveness of a spa residential program including physical activity (Sp-Ex) on bone cortical porosity compared with a spa residential program alone (Sp-alone) or physical activity alone (Ex-alone), in premenopausal women.
Variation of bone cortical porosity in premenopausal women | after 12 months
  To evaluate the effectiveness of a spa residential program including physical activity (Sp-Ex) on bone cortical porosity compared with a spa residential program alone (Sp-alone) or physical activity alone (Ex-alone), in premenopausal women.

SECONDARY OUTCOMES:
bone fracture risk | at Baseline, after 10 days, after 6 months, after 12 months
  questionnaire (FRAX - Fracture Risk Assessment Tool, bone fracture risks ; after registering results from DXA and personal details the computer calculates the fracture risks based on an algorithm)
General Health | at Baseline, after 10 days, after 6 months, after 12 months
  General Health will be measured using the General Health Questionnaire, (there is no score, just informative health information)
Greater short-term benefits on health factors with the Sp-Ex program than with Sp-alone or Ex-alone (Bone health will be obtained from the combination of 5 measures). | at Baseline, after 10 days, after 6 months, after 12 months
  Evaluate the effectiveness of the Sp-Ex program compared with the Sp-alone or Ex-alone on short-term modification of health factors among premenopausal women.
Physical Activity | at Baseline, after 10 days, after 6 months, after 12 months
  Quality of life will be measured using the SF-36 (Short Form 36 ; 9 sections questionnaire ; scale range from 0 (bad) to 100(excellent))
Quality of life | at Baseline, after 10 days, after 6 months, after 12 months
  Calcium intake will be measured using the Fardellonne questionnaire (recommended daily consummation in France: women 900 mg/d; women >55 years old 1200mg/d)
Calcium intake | at Baseline, after 10 days, after 6 months, after 12 months
  Depression and anxiety will be measured using Hamilton scale (scale range from 0 to 4, if > 20 high level of anxiety)
Depression and anxiety | at Baseline, after 10 days, after 6 months, after 12 months
  Depression and anxiety will be measured using the Hospital anxiety and depression scale (scale range from 0 to 3, with a total score between 0 to 21. Threshold score is 8)
Depression and anxiety | at Baseline, after 10 days, after 6 months, after 12 months
  anxiety will be measured using the state and trait anxiety inventory scale (scale range from 1 to 4, with a total score between 20 to 80. If <35 poor level of anxiety, if > 66 very high level of anxiety)
Anxiety | at Baseline, after 10 days, after 6 months, after 12 months
  Burn-out will be measured using the Maslach Burn Out Inventory (scale range from 0 to 6, with 0 = never and 6 = almost always)
Burn-out | at Baseline, after 10 days, after 6 months, after 12 months
  Job content will be measured using the Karasek questionnaire (scale range from 1 to 4, with 1= not agreed and 4 = totally agreed)
Job content | at Baseline, after 10 days, after 6 months, after 12 months
  Job content will be measured using the Karasek questionnaire (scale range from 1 to 4, with 1= not agreed and 4 = totally agreed)
Body mass | at Baseline, after 10 days, after 6 months, after 12 months
  Body mass (muscle and fat) will be measured using Impedancemeter
Anthropometry | at Baseline, after 10 days, after 6 months, after 12 months
  weight (kg) will be obtained according to the ISAK (International Society for the Advancement of Kinanthropometry) recommendations
Anthropometry | at Baseline, after 10 days, after 6 months, after 12 months
  height (m) will be obtained according to the ISAK (International Society for the Advancement of Kinanthropometry) recommendations
Anthropometry | at Baseline, after 10 days, after 6 months, after 12 months
  waist circumference (cm) will be obtained according to the ISAK (International Society for the Advancement of Kinanthropometry) recommendations
Basic biology | at Baseline, after 10 days, after 6 months, after 12 months
  HbA1c (mmol/mol) will be measured using endocrine assays
Basic biology | at Baseline, after 10 days, after 6 months, after 12 months
  HDLc (mmol/L) will be measured using endocrine assays
Basic biology | at Baseline, after 10 days, after 6 months, after 12 months
  LDL-cholesterol (mmol/L) will be measured using endocrine assays
Basic biology | at Baseline, after 10 days, after 6 months, after 12 months
  Triglyceride (TG-mmol/L) will be measured using endocrine assays
Vitamin D | at Baseline, after 10 days, after 6 months, after 12 months
  Vitamin D will be measured using endocrine assays
Leptin | at Baseline, after 10 days, after 6 months, after 12 months
  Leptin will be measured using endocrine assays
Pro-inflammatory cytokine | at Baseline, after 10 days, after 6 months, after 12 months
  Pro-inflammatory cytokine (IL-1β, IL-6, IL-1, TNFα, IFNγ) will be measured using endocrine assays
heart rate variability | at Baseline, after 10 days, after 6 months, after 12 months
  heart rate variability will be measured using Holter
electrodermal activity | at Baseline, after 10 days, after 6 months, after 12 months
  electrodermal activity (skin conductance) will be measured using Wirst band electrodes
physical activity behaviour | at Baseline, after 10 days, after 6 months, after 12 months
  physical activity behaviour will be measured using an activity journal (participant will have to write all their daily activity from when they wake up to when they go to bed)
physical activity behaviour | at Baseline, after 10 days, after 6 months, after 12 months
  will be measured using an accelerometer-pedometer watch (daily step count)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France